CLINICAL TRIAL: NCT07301125
Title: Myofunctional Therapy for Obstructive Sleep Apnea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ENT-2025-33821
Record Dates: First submitted 2025-11-25; First posted 2025-12-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Myofunctional Therapy; High-Resolution Manometry
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Myofunctional Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Myofunctional Therapy (Experimental): The intervention consists of 90 days of MFT (5-6 days/week) along with completing daily logs.
  MFT will include high-intensity swallowing exercises and respiratory muscle strength training.
  Before and after the MFT intervention period, there will be a research visit that includes answering questionnaires about symptoms and health, performing throat HRM, and assessing oral and facial muscles involved in swallowing.
  Interventions: Procedure: Myofunctional Therapy

INTERVENTIONS:
Procedure: Myofunctional Therapy — The intervention consists of 90 days of MFT (5-6 days/week) along with completing daily logs.
  MFT will include high-intensity swallowing exercises and respiratory muscle strength training.

SUMMARY:
The purpose of this study is to explore a new way to examine the function of the muscles using a technique called high-resolution manometry. The study will enroll 30 adults with OSA, all of whom will use the myofunctional therapy (MFT) devices for 3 months. High-resolution manometry will be used to measure the amount of pressure generated by the muscles of the throat when drinking water or breathing air, both with and without the MFT devices, and before and after the MFT intervention. If successful, this method can help us understand why sleep improves after MFT.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65
* New diagnosis of OSA (AHI ≥ 5) or failure of first-line OSA treatment
* Willingness to forego first-line OSA treatment or stop current OSA treatment for 3 months

Exclusion Criteria:

* Medical comorbidities that require restricting fluid intake (e.g., dysphagia, renal disease, liver disease, hyponatremia)
* Severe nasal obstruction
* Severe ankyloglossia
* Craniofacial abnormality
* Severe pulmonary disease
* Severe post-traumatic stress disorder (PCL-5 > 33)
* Very severe insomnia (ISI > 22)
* Body mass index (BMI) ≥30 kg/m2.
* History of TBI
* Known oropharyngeal or esophageal dysphagia
* Pregnancy
* Allergy to topical anesthetic
* Inability to fast for 6 hours
* Recent facial trauma
* Recent nasal, pharyngeal, laryngeal, or esophageal surgery
* Known nasal, pharyngeal or esophageal obstruction
* Current upper respiratory infection
* Insufficient internet/computer access to participate in remote study visit
* Severe excessive daytime sleepiness (risk of motor vehicle accidents)
* Heart failure, recent stroke, heart attack, etc.
* Nasal Obstruction Symptom Evaluation (NOSE) Scale >15

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
MFT treatment fidelity | Day 90
  Treatment fidelity of two common MFTs (high-intensity swallowing exercises, respiratory muscle strength training) in individuals with OSA. Treatment fidelity will be determined via measuring the percent of sessions completed relative to the targeted number of sessions.
Pressure generation in posterior upper airway musculature | Day 90
  Comparison of pressure generation in posterior upper airway musculature before and after MFT intervention as assessed with HRM

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Hoffmeister, PhD, CCC-SLP, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States